CLINICAL TRIAL: NCT02176499
Title: Natriuretic Effect of Telmisartan Versus Placebo in Patients With Mild-to-Moderate Hypertension On a Controlled Sodium Diet (100 mmol/Day)
Brief Title: Natriuretic Effect of Telmisartan Versus Placebo in Patients With Mild-to-Moderate Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 502.255
Record Dates: First submitted 2014-06-26; First posted 2014-06-27 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan

ARMS (3):
- Telmisartan, low dose (Experimental): 3 weeks placebo run-in (normal diet), 1 week placebo run-in (controlled sodium diet), 2 weeks double-blind treatment ,1 week placebo wash-out (controlled sodium diet)
  Interventions: Drug: Telmisartan, low dose; Drug: Placebo
- Telmisartan, high dose (Experimental): 3 weeks placebo run-in (normal diet), 1 week placebo run-in (controlled sodium diet), 2 weeks double-blind treatment, 1 week placebo wash-out (controlled sodium diet)
  Interventions: Drug: Telmisartan, high dose; Drug: Placebo
- Placebo (Placebo Comparator): 3 weeks placebo run-in (normal diet), 1 week placebo run-in (controlled sodium diet), 2 weeks double-blind treatment, 1 week placebo wash-out (controlled sodium diet)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Telmisartan, low dose
  Arms: Telmisartan, low dose
Drug: Telmisartan, high dose
  Arms: Telmisartan, high dose
Drug: Placebo

SUMMARY:
Study to compare the natriuretic effect of telmisartan to placebo in mild-to-moderate hypertensive patients on a controlled sodium diet as well as to explore the effects of telmisartan on norepinephrine, plasma renin activity (PRA), plasma aldosterone, urine potassium, creatinin, chloride, bicarbonate and uric acid excretion. Additionally it was assessed whether the natriuretic effect disappears after treatment when telmisartan is stopped. The effects of telmisartan on seated clinic blood pressure and the relationship between urine sodium loss and decrease in ambulatory blood pressure after the first dose were assessed descriptively. Assessment of safety was also considered.

ELIGIBILITY:
Inclusion Criteria:

* Mild-to-moderate hypertension as defined by a morning mean diastolic blood pressure from ≥ 90 and ≤ 115 mmHg and a mean systolic blood pressure ≤ 200 mmHg after five minutes in the seated position at the end of three weeks of placebo run-in treatment
* Male or female patients between 18 and 65 years of age, inclusive. Patients 60 to 65 years of age must have a screening 24-hour urine creatinine clearance rate of ≥ 1 mL/sec
* Ability to provide written informed consent

Exclusion Criteria:

* Pre-menopausal women (last menstruation ≤ one year to start of screening)
* Post-menopausal women (last menstruation > one year from start of screening or have had a hysterectomy and oophorectomy)

  * Who have < three months of stable estrogen replacement therapy at screening
  * Who will be on progesterone therapy at any time during the trial
* Known or suspected secondary hypertension
* Hepatic and/or renal dysfunction as defined by the following laboratory parameters:

  * ALT (alanine aminotransferase) or AST (aspartate aminotransferase) greater than two times the upper limit of reference range
  * Serum creatinine greater than 2.3 mg/dL
* Bilateral renal artery stenosis; renal artery stenosis in a solitary kidney; post-renal transplant
* NYHA (New York Heart Association) functional class CHF (chronic heart failure) III-IV
* Unstable angina, myocardial infarction or cardiac surgery within the preceding three months
* Stroke within the preceding six months
* PTCA (percutaneous transluminal coronary angioplasty) within the preceding three months
* History of angioedema
* Sustained ventricular tachycardia, atrial fibrillation, or other clinically relevant cardiac arrhythmias as determined by the clinical Investigator
* Hypertrophic obstructive cardiomyopathy, aortic stenosis, hemodynamically relevant stenosis of aortic or mitral valve
* Administration of digoxin or other digitalis-type drugs
* Patients with insulin-dependent and non-insulin-dependent diabetes mellitus
* History of drug or alcohol dependency
* Use of antihypertensive agents such as diuretics, ACE inhibitors, angiotensin II antagonists, α-blockers, β-blockers, calcium channel antagonists, direct vasodilators at any time during the trial
* Administration of other non-antihypertensive medications known to affect blood pressure (e.g., oral corticosteroids, MAO (monoamine oxidase) inhibitors, nitrates) at any time during the trial
* Chronic administration of high doses of NSAIDS and aspirin (e.g., ibuprofen for rheumatoid arthritis and osteoarthritis in total daily dose in excess of 1600 mg, aspirin in excess of 2 Gm per day)
* Chronic use of salt substitutes containing potassium chloride; potassium supplements; extreme dietary restrictions
* Clinically significant sodium depletion as defined by a serum sodium level less than 130 mEq/L
* Clinically significant hyperkalemia as defined by a serum potassium level greater than 6.0 mEq/L. Clinically significant hypokalemia as defined by a serum potassium level less than 3.0 mEq/L
* Patients receiving any investigational therapy within one month of signing the informed consent form. Note that patients who have participated in previous telmisartan studies may participate in this study provided there has been at least one month between discontinuing the previous study and signing the consent for the present study
* Known hypersensitivity to any component of telmisartan
* Any other clinical condition which, in the opinion of the principal Investigator, would not allow safe completion of the protocol and safe administration of trial medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 1999-02; Primary Completion 1999-07 (Actual)

PRIMARY OUTCOMES:
Cumulative urinary sodium loss | 0-4, 4-8, 8-24 hours post-dose at baseline, day 0, day 7 and 0-24 hours post-dose on days 1-6

SECONDARY OUTCOMES:
Cumulative urine sodium loss | 0-24 hours post-dose on days 8-13 and 0-4, 4-8, 8-24 hours post-dose on day 14
Changes in body weight | 24 hours post-dose on days -28, -21 to -14, -7, -1, 0, 7, 14 and 22
Changes in plasma norepinephrine | Baseline, on day 0 after the end of the 24 hour dosing interval, on days 7, 14 and 22
Changes in renin activity | Baseline, on day 0 after the end of the 24 hour dosing interval, on days 7, 14 and 22
Changes in aldosterone | Baseline, on day 0 after the end of the 24 hour dosing interval, on days 7, 14 and 22
Changes in urine potassium | Baseline, on day 0 after the end of the 24 hour dosing interval, on days 7, 14 and 22
Changes in creatinine chloride | Baseline, on day 0 after the end of the 24 hour dosing interval, on days 7, 14 and 22
Changes in bicarbonate | Baseline, on day 0 after the end of the 24 hour dosing interval, on days 7, 14 and 22
Changes in uric acid | Baseline, on day 0 after the end of the 24 hour dosing interval, on days 7, 14 and 22
Cumulative urinary sodium gain during wash-out period | 0-24 hours post-dose on days from day 15 to 22
Changes in seated clinic blood pressure | Baseline and day 14
Changes in 24 hour ambulatory Blood Pressure (ABPM) after the first dose of telmisartan | Day 0
Number of patients with adverse events | up to 50 days
Number of patients with abnormal findings in physical examination | Baseline and day 22
Number of patients with abnormal findings in 12-lead electrocardiogram (ECG) | Baseline and day 22
Number of patients with abnormal changes in laboratory parameters | Baseline and day 22